CLINICAL TRIAL: NCT04976036
Title: Phase II Monocentric Randomized Study on Efficacy of Nintedanib for Treatment of Epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT) Patients
Brief Title: Efficacy of Nintedanib for Treatment of Epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT) Patients
Acronym: EPISTOP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Romain Lazor (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Dr. Romain Lazor, Head of interstitial and rare lung disease Unit, Principal investigator, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1199-0433
Record Dates: First submitted 2021-04-10; First posted 2021-07-26 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
Keywords: nintedanib; epistaxis; treatment
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nintedanib (Experimental): nintedanib 150 mg once a day for 2 weeks, then twice a day for 14 weeks
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator): placebo 150 mg once a day for 2 weeks, then twice a day for 14 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib — 150 mg oral nintedanib soft caps, once a day for 2 weeks and twice a day for 10 weeks (12 hours interval)
  Arms: Nintedanib
Drug: Placebo — 150 mg oral placebo soft caps, once a day for 2 weeks and twice a day for 10 weeks (12 hours interval)
  Arms: Placebo

SUMMARY:
Patients affected by hereditary hemorrhagic telangiectasia (HHT) very often suffer from recurrent nosebleeds called epistaxis. There is no treatment currently available to reduce the frequency or severity of epistaxis.

This research project will examine the effect of nintedanib, a capsule to be taken twice a day, on the frequency and severity of epistaxis in HHT.

The study will take place at the Respiratory medicine department of the Lausanne University Hospital (Centre hospitalier universitaire vaudois, CHUV). The investigators will recruit about 48 participants with HHT, who will be divided in 2 groups. Each group will perform the same examinations and follow-up visits. The study will begin with 2 months of observation during which subjects will be asked to fill a diary to record the number and duration of epistaxis episodes. The diary will be filled daily for the entire duration of the study, i.e. 8 months. After 2 months of observation, the treatment phase will begin. Participants will take a capsule (nintedanib 150 mg or placebo) once a day for 2 weeks, then twice a day for 14 weeks. In case of intolerance at the dose of 2 capsules per day, the treatment may be reduced to 1 capsule per day. Subjects will also have to mention on the diary any blood transfusion, iron perfusion, and any symptoms they may be experiencing. Following the 16 weeks of treatment, an 8-week follow-up period will allow to observe the effects of nintedanib after the end of the treatment period, and to monitor any unexpected adverse events.

DETAILED DESCRIPTION:
Hereditary hemorrhagic telangiectasia (HHT), or Rendu-Osler-Weber disease, is a rare genetic disease with autosomal dominant transmission and a prevalence in the general population of 1/5'000 to 1/10'000. Genetic mutations in HHT affect the intracellular angiogenic signalling pathways (for example through the Vascular Endothelial Grow Factor [VEGF]) in endothelial cells. Clinically, HHT leads to arteriovenous malformations in various organs including the lung, brain, liver, digestive tract, skin, and nasal mucosa. More than 90% of HHT patients suffer from chronic nosebleeds called epistaxis, which may lead to severe iron deficiency, anemia requiring recurrent blood transfusions in 10-30%, emergency hospital admissions for acute and sometimes life-threatening bleeding, and moderate to severe reduction in quality of life in about 70%. Nintedanib, an antifibrotic drug approved for the treatment of idiopathic pulmonary fibrosis (IPF), also targets the VEGF receptor. The investigators hypothesize that nintedanib, acting by inhibition of the VEGF receptor, may reduce the duration and frequency of epistaxis in HHT patients.

This hypothesis will be studies in a phase II randomized controlled trial. The study design will be the following:

Pre-therapeutic observation period of 8 weeks followed by a 16-week interventional phase (nintedanib 150 mg once a day for 2 weeks, then twice a day for 14 weeks compared to a placebo at same regimen), and by an 8-week follow-up period to assess post-treatment effects and possible adverse events.

Number of randomized patients: up to 24 in each arm, to achieve at least 16 patients completing the entire study in each arm, with up to 8 drop-out in each arm allowed.

Patients will complete an epistaxis self-administered assessment grid daily since the screening visit, and an epistaxis severity score and a quality of life assessment at the end of weeks 8, 16, 20, 24 and 32.

Blood will be sampled at screening (= week 1), and at weeks 8, 12, 16, 20, 24 and 32 to assess hemoglobin and ferritin levels, and to monitor hepatic or renal functions for safety reasons.

Microphotography (dermoscopy) of selected cutaneous telangiectasia will be performed at visits 1, 6 and 7.

Prior to study initiation, the study protocol, the patient information form and consent form, as well as other study-specific documents will be submitted to the local ethics committee (CER-VD) and the Swiss national drug regulatory authority (Swissmedic) for approval. Any amendment to the protocol must be approved (if legally required) by these institutions.

Participants will be closely monitored for adverse events at each visit. Each participant will hold of an emergency card indicating his/her randomization number, the name and number of the study, the name of the PI, the possible Investigated Medical Product (IMP) i.e. nintedanib or placebo, and the emergency phone number. In case of serious adverse event (SAE), participants may call the emergency number. The call will be answered directly by the PI or a co-investigator.

Individual medical information obtained during the course of this study will be confidential and disclosure to third parties will be prohibited. Confidentiality will also be warranted by using coded subject identification in the computer files.

Only authorized staff of the research team, i.e. the sponsor-PI, investigators, and study nurse will be authorized to access participants data in a password-protected database. After database lock, the Sponsor-PI, investigators and statistician will be able to access the database for analysis. The database will be archived for ten years after study completion.

ELIGIBILITY:
Inclusion criteria:

1. signed informed consent
2. definite HHT disease (defined as the presence of a pathogenic mutation in one of the HHT genes, or the presence of 3 out of 4 Curaçao clinical criteria)
3. age ≥18 years at the time of informed consent
4. moderate to serious epistaxis defined as Epistaxis Severity Score (ESS) ≥2.5
5. absence of cerebral arteriovenous malformation demonstrated by brain imaging

Exclusion criteria:

1. Women who are pregnant or breastfeeding
2. For women of childbearing potential (WOCBP, see Annex VII for definition), non-agreement to follow instructions for method(s) of contraception for the heterosexual couple (see Annex VII for instructions) during the treatment period and follow-up, or at least 3 months after the last dose of IMP, or if there are concerns that they will not reliably comply with the contraception requirements.
3. Acute infection
4. aspartate aminotransferase (AST), or alanine aminotransferase (ALT), or total bilirubin >1.5x (or >2.5x in patients known for Gilbert's syndrome) the upper limit of normal
5. Renal clearance by Cockcroft-Gault formula <30 ml/min
6. Untreated pulmonary arteriovenous malformation (if vaso-occlusion is technically feasible)
7. Hemoptysis or hematuria within the last 12 months
8. Ulcus or active gastric bleeding within the last 12 months
9. Anticoagulant or antiplatelets treatment
10. Coronary heart disease
11. Thrombotic event within the last 12 months
12. Long QT syndrome (on ECG performed at screening)
13. Known allergy to nintedanib, soya, peanuts
14. Bevacizumab, pazopanib or other anti-angiogenic treatments within the last 12 months
15. Concomitant treatment with ketoconazole, erythromycin, rifampicin, carbamazepine, phenytoin, St John's Wort
16. Surgery within the last 3 months or planned within the next 9 months
17. Recent unhealed wound
18. Any other serious underlying medical condition that could interfere with the study treatment and potential adverse events
19. Any mental or other impairment that may compromise compliance with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change of epistaxis duration in minutes under nintedanib treatment as compared to placebo in HHT patients. | Week 0 to week 7
  The primary outcome will be the proportion of patients with at least 30% change of monthly epistaxis duration in minutes after 16 weeks of study treatment (at V6, week 24) compared to baseline (V1, week 8) assessed in nintedanib arm and in placebo arm.
  * The monthly epistaxis duration after 16 weeks of study treatment is defined as the average of epistaxis duration during the last 12 weeks of study treatment (minutes/4-weeks period averaged for weeks 12 to 24, i.e. V3 to V6)
  * The monthly epistaxis duration at baseline is defined as the average of epistaxis duration during the observation period (minutes/4-weeks period averaged for weeks 1 to 8, i.e. V0 to V1).

SECONDARY OUTCOMES:
Change in number of epistaxis episodes per 4 weeks | Secondary endpoints will be evaluated at week 8, 16, 20, 24 and 32
  Number of epistaxis will be recorded daily by participants on the daily grid and the number of episodes per 4 weeks will be compared between baseline and treatment period at V3-V6
Change in the Nasal Outcome for Epistaxis in Hereditary Hemorrhagic Telangiectasia score | Secondary endpoints will be evaluated at week 8, 16, 20, 24 and 32
  The Nasal Outcome for Epistaxis in Hereditary Hemorrhagic Telangiectasia (NOSE HHT questionnaire) wil be used to measure physical, social and emotional impacts of epistaxis. It is a 29-items questionnaire using a Likert scale. A higher score indicates a worse outcome. Comparison will be made between the observation period and the treatment period and follow-up.
Change in number of blood transfusions per 4 weeks | Secondary endpoints will be evaluated at week 8, 12, 16, 20, 24 and 32
  Participants will record number of blood transfusions on the daily grid. Comparison will be made between the observation period and the treatment period and follow-up.
Change in epistaxis severity score (ESS) | Secondary endpoints will be evaluated at week 8, 16, 24 and 32
  Epistaxis Severity Score (ESS) is a 6-item score. Each answer gives a number of points which is multiplied by a coefficient. The sum of the 6 answers provides the score. A higher score indicates a worse outcome. The score during the observation period will be compared to the score during the treatment period and follow-up.
Change in number of iron infusions per 4 weeks | Secondary endpoints will be evaluated at week 8, 12, 16, 20, 24 and 32
  Participants will record the number of iron perfusions on the daily grid. Comparison will be made between the observation period and the treatment period and follow-up.
Change in hemoglobin level in g/l | Secondary endpoints will be evaluated at week 8, 12, 16, 20, 24 and 32
  Comparison will be made between the observation period and the treatment period and follow-up.
Change in ferritin level in ng/ml | Secondary endpoints will be evaluated at week 8, 12, 16, 20, 24 and 32
  Comparison will be made between the observation period and the treatment period and follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory medicine Department, Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data are available on request.

REFERENCES:
- [Background] Robert F, Desroches-Castan A, Bailly S, Dupuis-Girod S, Feige JJ. Future treatments for hereditary hemorrhagic telangiectasia. Orphanet J Rare Dis. 2020 Jan 7;15(1):4. doi: 10.1186/s13023-019-1281-4. PMID 31910860
- [Background] Kovacs-Sipos E, Holzmann D, Scherer T, Soyka MB. Nintedanib as a novel treatment option in hereditary haemorrhagic telangiectasia. BMJ Case Rep. 2017 Jun 26;2017:bcr2017219393. doi: 10.1136/bcr-2017-219393. PMID 28652319